CLINICAL TRIAL: NCT06330363
Title: The Impact of Low Level Laser Treatment on Skeletal Muscle and Skin Tissue Mitochondrial Respiration, Metabolic Activity and Signalling in Vivo in Humans
Brief Title: The Impact of Low Level Laser Treatment on Skeletal Muscle and Skin Tissue
Acronym: LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: METC 23-049
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Muscles Metabolism; Skin Metabolism
MeSH Terms: interventions — Laser Therapy; salicylhydroxamic acid; Light

STUDY DESIGN:
Intervention Model Description: Within-subject study
Who Masked: Participant, Outcomes Assessor
Masking Description: One let will receive the laser therapy, the other one will get a sham laser. The person analyzing the samples will be blinded to legs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLLT (Experimental): The LLLT will be performed using a Cube plus30 (Eltech K-Laser s.r.l., Italy). Settings will be based on manufacturer's guidelines for skin and deep tissue stimulation. The LLLT will take 25 min, with 3x5 min of treatment separated by 5 min of rest. In total 16800 J in form of light energy will be applied (3 x 5600 J). All 4 available wavelength will be used (660, 800, 905 and 970 nm). The randomization procedure to allocate the treated leg will occur via a random-number generator stratified for sex (www.randomization.com) performed by an independent researcher of the research group. During the laser treatment protective goggles (K-Laser Protective Goggles, Eltech K-Laser s.r.l.) need to be worn and will therefore be provided. LLLT will only be applied by trained personal.
  Interventions: Other: Laser therapy
- Sham (Sham Comparator): Sham laser based on the same laser device which emitts only light.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Laser therapy — The Cube plus30 from Eltech K-Laser s.r.l. (Italy, www.k-laser.com) will be used for LLLT. The laser devices from Eltech K-Laser s.r.l. have been used in (clinical) studies with a variety in patient populations (38-41) and clinical practice (https://resources.k-laser.com.au/medical-laser-clinical-applications). The device is a registered medical device in the EU confirmed by Kiwa Cermet Italia.
  Arms: LLLT
Other: Sham — The laser device has sham light option that will be used.
  Other Names: Light
  Arms: Sham

SUMMARY:
Rationale: Low level laser therapy, or photobiomodulation, is getting more attention as a non-invasive treatment strategy for numerous conditions. Phototherapy has been applied for more than 40 years for the treatment of musculoskeletal and neurological conditions. Low level laser therapy generally applies red or near-infrared lasers with a wavelength between 600 and 1000 nm and low power wattage from 5 to 500 mW and a power density between 1 and 5 W/cm2. The laser light is absorbed by the skin without thermal damage and penetrates deeply into tissues where it is supposed to induce its physiological effects at the cellular level. Laser therapy has been hypothesized to stimulate mitochondrial respiration, increase tissue oxygenation, and support tissue regeneration. Despite supportive research data on in vitro cell and in vivo animal data, there are surprisingly few data on the proposed impact of low level laser treatment (LLLT) on tissue metabolism in vivo in humans.

Objective: To assess the impact of acute laser treatment on muscle tissue mitochondrial respiration in vivo in healthy, young adults. Secondary objectives include the in vivo assessment of cellular energy, anabolic, angiogenic and inflammatory pathways, along with enzyme activity within muscle and skin.

Study design: Within-subject study.

Study population: 12 healthy (BMI 18.5-30 kg/m2) young (age: 18-35 y) adults (6 men and 6 women).

Intervention: One leg of the subjects will receive LLLT, while the other leg will receive no treatment. After the treatment muscle and skin biopsy samples will be taken from both legs.

Main study parameters/endpoints: The primary outcome will be mitochondrial respiration of the LLLT treated and non-treated leg based on muscle samples. Secondary study parameters are muscle and skin gene expression, protein signalling and enzyme activity.

DETAILED DESCRIPTION:
The present study utilizes an acute within-subject design in healthy young adult participants. In total, 12 healthy young adults (6 men and 6 women) will participate in the study. Participants' legs will be randomly assigned to low level laser treatment or no treatment (Figure 1). Each participant will participate in a screening session (~1 h) and 1 experimental test day (~1.5 h). Figure 1 shows a graphical illustration of the study overview.

In total, 12 healthy (BMI 18.5-30 kg/m2) young (age: 18-35 y) males and females will participate in the present study. The nature and the risks of the experimental procedures will be explained to all subjects before their informed consent will be obtained. All subjects will be recruited through social media and advertisements on dedicated bulletin boards within the MUMC+ buildings and local shops will be used.

Each subject will participate in an experimental trial lasting ~1.5 h. Subjects will be instructed to arrive at the university at 9:00 AM in an overnight fasted and rested state, meaning that participants are not allowed to eat and drink (except for water) from 21:00 the night prior to the experimental trial. They will be instructed to come to the university by car or public transportation. After the subjects arrive at the University, we will ask them to put on their shorts, determine their body mass, and assign them to a bed. Subjects will rest in a supine position for 10 minutes. Thereafter, the LLLT will be applied on one leg, which will be randomized. The other leg will receive no treatment. Immediately after the treatment muscle biopsies will be taken from the m. vastus lateralis of both legs. The muscle biopsy from the treated leg will be sampled 15 min after finishing the LLLT. Additionally, skin biopsies will be taken from the same area. The skin biopsy of the treated leg will be collected 20 min after finishing the LTT. During the test day, a total of 2 muscle and skin biopsies will be taken, 1 biopsy from each leg. Here each skin biopsy sampling consists of 2 4 mm punch biopsies. The time between finishing the LLLT and collection of the tissue samples will be noted.

Primary objective: To assess the impact of acute laser treatment on muscle tissue mitochondrial respiration in vivo in healthy, young adults.

Secondary objective: To assess the impact of acute laser treatment on muscle cellular energy, anabolic, angiogenic and inflammatory pathways, along with enzyme activity.

Tertiary objectives: To assess the impact of acute laser treatment on skin cellular energy, anabolic, angiogenic and inflammatory pathways, along with enzyme activity.

Hypothesis:

1. It is hypothesized that muscle mitochondrial respiration will be higher following low level laser treatment.
2. It is hypothesized that muscle gene expression, protein signalling and enzyme activity will be higher following low level laser treatment.
3. It is hypothesized that skin gene expression, protein signalling and enzyme activity will be higher following low level laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* Aged between 18 and 35 y inclusive
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Participating in a structured (progressive) exercise program or >4h of vigorous physical activity per week.
* Smoking regularly (i.e. >5 cigarettes/week)
* Pregnancy
* Hormonal replacement therapy
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g. diabetes)
* Diagnosed skin disorders
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of anti-coagulants

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Muscle mitochondrial respiration | only one time point, immediately after the intervention
  Maximal complex I+II-linked mitochondrial respiration of muscle tissue, expressed as oxygen consumption (JO2) in units of pmol/sec/mg dry weight muscle. Oxygen consumption will be monitored in an Oroboros O2K Oxygraph (Innsbruck, Austria) in the presence of pyruvate, malate, ADP, glutamate, and succinate, providing substrates to maximally stimulate complex I+II-linked respiration.

SECONDARY OUTCOMES:
Gene expression (mRNA) via real-time PCR | only one time point, immediately after the intervention
  of muscle and skin
Protein expression via western blotting | only one time point, immediately after the intervention
  of muscle and skin
Skin mitochondrial respiration | only one time point, immediately after the intervention
  Maximal complex I+II-linked mitochondrial respiration of skin tissue, expressed as oxygen consumption (JO2) in units of pmol/sec/mg dry weight muscle. Oxygen consumption will be monitored in an Oroboros O2K Oxygraph (Innsbruck, Austria) in the presence of pyruvate, malate, ADP, glutamate, and succinate, providing substrates to maximally stimulate complex I+II-linked respiration.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided